CLINICAL TRIAL: NCT04883515
Title: Effects of Oral Glutamine Supplementation on Insulin Resistance and Functional Intestinal Disorders in Obese Patients.
Acronym: OBEGLUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/0334/HP
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Insulin Resistance
Keywords: oral glutamine supplementation
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral glutamine supplementation (Experimental): patient will receive Oral glutamine supplementation 10 g Ter In Die during 8 weeks
  Interventions: Dietary Supplement: Oral glutamine supplementation; Procedure: Insulin-resistance evaluation; Procedure: Functional intestinal disorders evaluation
- Oral protein powder supplementation (Active Comparator): patient will receive Oral protein powder supplementation10 g Ter In Die during 8 weeks
  Interventions: Dietary Supplement: Oral protein powder supplementation; Procedure: Insulin-resistance evaluation; Procedure: Functional intestinal disorders evaluation

INTERVENTIONS:
Dietary Supplement: Oral glutamine supplementation — patient will receive oral glutamine supplementation 10 g Ter In Die during 8 weeks
  Arms: Oral glutamine supplementation
Dietary Supplement: Oral protein powder supplementation — patient will receive oral protein powder supplementation10 g Ter In Die during 8 weeks
  Arms: Oral protein powder supplementation
Procedure: Insulin-resistance evaluation — Homeostasic model assessment of insulin resistance test will be performed at baseline, Week 8 and Week 16
Procedure: Functional intestinal disorders evaluation — Functional intestinal disorders will be measured by the IBS severity score and feces consistency by Bristol scale at baseline, Week 8 and Week 16

SUMMARY:
Obesity, which has a prevalence at 15% in France, is a major public health concern. Altered glycemic control and irritable bowel syndrome (IBS) are frequently observed in obese patients and lead to reduce the quality of life. In the last decades, the role of gut microbiota and intestinal permeability has been underlined in obesity, glycemic control and IBS. Interestingly, experimental and clinical data show that glutamine, an amino acid, is able to maintain or restore intestinal permeability in different conditions. We thus hypothesize that oral glutamine supplementation may restore gut barrier function contributing to improve glycemic control and IBS-symptoms. Our project will thus aim to evaluate the effects of 8 weeks - oral glutamine supplementation on glycemic control and IBS symptoms in obese patients in a blinded randomized controlled trial. Placebo group will received protein powder. 55 obese patients will enrolled in each arm and will received oral glutamine supplementation or protein powder (10g t.i.d.) during 8 weeks. Blood and feces samples and intestinal permeability assays will be performed at baseline (w0), after 8 weeks of supplementation (w8) and then after 8 weeks of a wash-out period (w16).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 65 years
* Patient with h grade II or III obesity (body mass index equal or higher than 35 kg/m2)
* Patient with insulino-resistance (fasting glycaemia ≥ 1g/l et < 1.26 g/l)
* Patient with irritable bowel syndrome (Rome IV criteria ≥ 2)

Exclusion Criteria:

* Patient with Known liver insufficiency (prothrombin time < 70%)
* Patient with Known kidney failure (GFR < 60 ml/mn)
* Patient with Known intestinal diseases such as inflammatory bowel diseases
* Vomiting patients (≥ 1/ day) during the last 4 weeks
* Patient Previously received bariatric surgery or digestive surgery
* Patient Using laxatives or protein powder during the 4 last weeks
* On going Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change between Homeostasic model assessment of insulin resistance test value at baseline and week 8 | Week 8

SECONDARY OUTCOMES:
Change between Homeostasic model assessment of insulin resistance test value at baseline and week 16 | Week 16
Change between Homeostasic model assessment of insulin resistance test value at Week 8 and week 16 | week 16
Change between Irritable Bowel Syndrome (IBS) severity score at baseline and week 8 | Week 8
  Francis score will be used
Change between Irritable Bowel Syndrome (IBS) severity score at baseline and week 16 | Week 16
  Francis score will be used
Change between feces consistency at baseline and week 8 | Week 8
  bristol scale will be used
Change between feces consistency at baseline and week 16 | Week 16
  bristol scale will be used

CONTACTS AND LOCATIONS:
Overall Officials: Hélène LELANDAIS, MD, Principal Investigator — University Hospital, Rouen; Moïse COEFFIER, Pr, Study Director — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No